CLINICAL TRIAL: NCT02416076
Title: Evaluation of the Ulthera® System for Lifting and Tightening the Face and Neck Using Standard Transducers Versus Simulines Transducers
Brief Title: Ultherapy® for Treating the Face and Neck Using Standard Versus Simulines Transducers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-141
Record Dates: First submitted 2015-02-26; First posted 2015-04-14 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2016-02

CONDITIONS: Skin Laxity
Keywords: Ulthera® System; Ultherapy®; Ulthera, Inc.
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Group A - LT side simulines Ulthera treatment at EL2 (Active Comparator): Ulthera treatment using 'Ulthera System, prototype simulines transducers' on the LEFT side of the face and 'Ulthera System, standard transducers' on the RIGHT of the face at the default Energy Level [EL2].
  Interventions: Device: Ulthera Treatment at EL2
- Group B - RT side simulines Ulthera treatment at EL2 (Active Comparator): Ulthera treatment using 'Ulthera System, prototype simulines transducers' on the RIGHT side of the face and 'Ulthera System, standard transducers' on the LEFT side of the face at the default Energy Level [EL2] .
  Interventions: Device: Ulthera Treatment at EL2
- Group C - LT side simulines Ulthera treatment at EL4 (Active Comparator): Ulthera treatment using 'Ulthera System, prototype simulines transducers' on the LEFT side of the face and 'Ulthera System, standard transducers' on the RIGHT of the face at a higher Energy Level [EL4].
  Interventions: Device: Ulthera Treatment at EL4
- Group D - RT side simulines Ulthera treatment at EL4 (Active Comparator): Ulthera treatment using 'Ulthera System, prototype simulines transducers' on the RIGHT side of the face and 'Ulthera System, standard transducers' on the LEFT side of the face at a higher Energy Level [EL4] .
  Interventions: Device: Ulthera Treatment at EL4
- Group E - LT side simulines/standard Ulthera treatment at EL4 (Active Comparator): Ulthera treatment using a 4-4.5 'Ulthera System, prototype simulines transducers' and 7-3.0 'Ulthera System, standard transducers' on the LEFT side of the face and 'Ulthera System, standard transducers' on the RIGHT of the face at a higher Energy Level [EL4].
  Interventions: Device: Ulthera Treatment at EL4
- Group F - RT side simulines/standard Ulthera treatment at EL4 (Active Comparator): Ulthera treatment using a 4-4.5 'Ulthera System, prototype simulines transducers'and 7-3.0 standard transducer on the RIGHT side of the face and 'Ulthera System, standard transducers' on the LEFTof the face at a higher Energy Level [EL4].
  Interventions: Device: Ulthera Treatment at EL4

INTERVENTIONS:
Device: Ulthera Treatment at EL2 — Focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ultherapy
  Arms: Group A - LT side simulines Ulthera treatment at EL2; Group B - RT side simulines Ulthera treatment at EL2
Device: Ulthera Treatment at EL4 — Focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ultherapy
  Arms: Group C - LT side simulines Ulthera treatment at EL4; Group D - RT side simulines Ulthera treatment at EL4; Group E - LT side simulines/standard Ulthera treatment at EL4; Group F - RT side simulines/standard Ulthera treatment at EL4

SUMMARY:
Up to 40 participants will be enrolled, randomized and treated. Enrolled participants will receive one, split-face Ulthera® treatment on the face and neck using a Ulthera System standard transducer on one side of the face and a Ulthera System prototype simulines transducers on the other side of the face. Follow-up visits will occur at 90 and 180 days post-treatment. Study images will be obtained pre-treatment, immediately post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This is a prospective, multi-center, split-face, randomized pilot trial to determine the clinical feasibility of the Ulthera System prototype simulines transducers, that is, transducers which deliver two lines of treatment simultaneously (at once), in comparison to the standard transducers which deliver a single treatment line, by collecting average pain scores in the treated regions, as well as efficacy and treatment efficiency data. There will be 3 study arms with each arm having 2 treatment groups. Enrolled participants will be randomized to one of two study arms, and one of two treatment groups within each study arm.to determine which side of the face will be treated with Ulthera System standard transducers and Ulthera System prototype simulines transducers and the energy level for treatment. Participants will receive one dual-depth treatment at 4.5 millimeter (mm) and 3.0mm depths.

Clinical feasibility will be assessed based on comfort level of standard transducers versus simulines transducers by comparing average pain scores obtained during study treatment. Efficacy will be determined based on qualitative masked assessment of post-treatment photographs compared to pre-treatment photographs and quantitative eyebrow lift measurements. Patient satisfaction questionnaires will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 30 to 65 years.
* Participant in good health.
* Skin laxity on the area(s) to be treated.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Participants of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control (example barrier methods used with a spermicidal agent, hormonal methods, intrauterine device (IUD), surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

  1. Postmenopausal for at least 12 months prior to study;
  2. Without a uterus and/or both ovaries; or
  3. Bilateral tubal ligation at least six months prior to study enrollment.
* Absence of physical or psychological conditions unacceptable to the investigator.
* Willingness to refrain from use of aspirin, Ibuprofen, Naproxen or any other nonsteroidal anti-inflammatory drug (NSAID) prior to each study treatment and chronic use during the entire posttreatment study period. Washout period, if chronic user, for 4 weeks prior to the first treatment. Washout period for limited acute NSAID use, that is, a maximum of 2-3 doses, is required in the 2 weeks prior to any study treatment visit.
* Willingness and ability to provide written consent for study-required photography and adherence to photography procedures (that is, removal of jewelry and makeup).
* Willingness and ability to provide written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization prior to performance of any study-related procedure.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Excessive subcutaneous fat in the area(s) to be treated.
* Excessive skin laxity on the area(s) to be treated.
* Significant scarring in the area(s) to be treated.
* Open wounds or lesions in the area(s) to be treated.
* Severe or cystic acne on the area(s) to be treated.
* Active implants (example, pacemakers or defibrillators), or metallic implants in the treatment areas (dental implants not included).
* Inability to understand the protocol or to give informed consent.
* Microdermabrasion, or prescription level glycolic acid treatment to the treatment area(s) within two weeks prior to study participation or during the study.
* Marked asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area(s) to be treated.
* BMI equal to or greater than 25.
* History of chronic drug or alcohol abuse.
* History of autoimmune disease.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
* Participants who anticipate the need for surgery or overnight hospitalization during the study.
* Participants who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
* Concurrent enrollment in any study involving the use of investigational devices or drugs.
* Current smoker or history of smoking in the last five years.
* Current user of any nicotine-containing products, example, electronic cigarettes (e-cigarettes), Nicorette gum, nicotine patches, etc.
* History of the following cosmetic treatments in the area(s) to be treated:

  1. Skin tightening procedure within the past year;
  2. Injectable filler of any type within the past:

  i.12 months for Hyaluronic acid fillers (example Rstylane)

ii.12 months for Ca Hydroxyapatite fillers (example Radiesse)

iii. 24 months for Poly-L-Lactic acid fillers (example Sculptra)

iv. Ever for permanent fillers (example Silicone, ArteFill)

c. Neurotoxins within the past six months; d. Ablative resurfacing laser treatment; e. Nonablative, rejuvenative laser or light treatment within the past six months; f. Surgical dermabrasion or deep facial peels; g. Facelifts, blepharoplasty, or browlift within the past 18 months; or h. Any history of contour threads.

* History of using the following prescription medications:

  1. Accutane or other systemic retinoids within the past six months;
  2. Topical Retinoids within the past two weeks;
  3. Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix);
  4. Psychiatric drugs that in the investigators opinion would impair the participant from understanding the protocol requirements or understanding and signing the informed consent.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2015-09-23 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Comfort level of standard transducers versus simulines transducers during Ultherapy® treatment | During study treatment. Participants will be followed for an average of 90 minutes.
  Subjects' treatment-related pain scores will be obtained using a validated 0-10 point Numeric Rating Scale while study treatment is being administered. It is estimated that each study treatment will be completed in approximately 90 minutes.

SECONDARY OUTCOMES:
Brow lift obtained using simulines versus standard transducers | 90 days post-treatment
  Brow lift as assessed by quantitative measurements of pre- to post-treatment photos.
Brow lift obtained using simulines versus standard transducers | 180 days post-treatment
  Brow lift as assessed by quantitative measurements of pre- to post-treatment photos.
Improvement in overall lifting and tightening of skin | 90 days post-treatment
  As assessed by a masked, qualitative assessment of photographs at 90 days post-treatment compared to baseline.
Improvement in overall lifting and tightening of skin | 180 days post-treatment
  As assessed by a masked, qualitative assessment of photographs at 180 days post-treatment compared to baseline.
Patient Satisfaction | 90 days post-treatment
  As assessed by a patient satisfaction questionnaire completed by the subject.
Efficiency of simulines versus standard transducers | During study treatment
  As determined by comparing treatment times using the simulines transducers compared to treatment times using the standard transducers.

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (3):
- United States (3):
  - Clinical Testing of Beverly Hills, Beverly Hills, California
  - California Skin Institute - Saratoga, Saratoga, California
  - Wilmington Dermatology Center, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: No